CLINICAL TRIAL: NCT00558038
Title: Comparison of Different Treatment Regimens in Patients With Stage 1-2 Type C Hepatic Encephalopathy: AST-120 vs Lactulose
Brief Title: Safety and Efficacy of AST-120 Compared to Lactulose in Patients With Hepatic Encephalopathy
Acronym: AST015
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocera Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AST015
Record Dates: First submitted 2007-11-09; First posted 2007-11-14 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic; Encephalopathy; Liver; Liver Disease; Liver Failure; Lactulose; AST-120
MeSH Terms: conditions — Hepatic Encephalopathy; Brain Diseases; Liver Diseases; Liver Failure | interventions — AST 120; Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: lactulose
- 2 (Experimental)
  Interventions: Drug: AST-120

INTERVENTIONS:
Drug: AST-120 — AST-120
  Arms: 2
Drug: lactulose — lactulose
  Other Names: Chronulac, Constilac, Constulose, Duphalac, Evalose
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the experimental drug AST-120 compared to lactulose in patients with mild hepatic encephalopathy.

DETAILED DESCRIPTION:
This is a multi-center, open-label, four week trial comparing AST-120 to lactulose in patients with mild (Stage 1-2) hepatic encephalopathy.

Patients will be randomized into two groups:

* Lactulose
* AST-120

Patients meeting the inclusion criteria will take either AST-120 or lactulose for 4 weeks (28 days). AST-120 will be distributed in 2 gram sachets to be taken four times daily. Lactulose will be taken in the same formulation, at the same dose and frequency as previously prescribed for the individual patient.

Lactulose naïve patients who are randomized to lactulose will receive an initial dose of 30cc twice a day. The dose should be titrated at the discretion of the investigator until the patient is experiencing 2-3 soft stools per day.

Patients randomized to AST-120 will receive 2 grams four times a day for the duration of the study. Titration of AST-120 will NOT be allowed.

Patients will be evaluated throughout the study for efficacy and safety. A follow-up visit will be scheduled 1 week after the end of the 4 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with End Stage Liver Disease secondary to any cause (patients who have undergone portosystemic shunting (TIPS) procedure > 3 months prior to randomization can be included)
* Lactulose naïve patients or patients currently on an established dose of lactulose
* MELD score ≤ 15 (MELD score up to 20 is allowable if it has remained stable for at least 3 months)
* Meet the criteria for Stage 1-2 hepatic encephalopathy according to the Westhaven Scale
* Patients must have discontinued rifaximin or other oral antibiotics for at least 48 hours prior to randomization
* Able and willing to comply with all protocol procedures for the planned duration of the study
* Able and willing to understand, sign and date an informed consent document, and authorize access to protected health information
* Have a person (spouse, relative, or friend) willing to accompany the patient to the study visits (patients in this condition are not recommended to drive a vehicle)
* Females must be postmenopausal, surgically incapable of bearing children, or practicing a reliable method of birth control (intrauterine devices, spermicide and barrier). Partner/spouse sterility may also qualify at the investigator's discretion. Females of child-bearing potential must have a negative urine pregnancy test at baseline.

Note: Patients already on lactulose and randomized to AST-120 will stop taking lactulose on the day they begin taking AST-120.

Exclusion Criteria:

* Patients whose condition necessitates continuous administration of antibiotics (e.g. rifaximin, neomycin, metronidazole)
* Patients undergoing chemotherapy for treatment of cancer (patients with hepatocellular carcinoma being treated by methods other than chemotherapy may be enrolled)
* Patients who require continued treatment with narcotics or sedatives
* Patients who have active GI bleeding
* Patients who have an active infection
* Patients who have signs and symptoms of severe dehydration
* Poor tolerability of venipuncture or lack of adequate venous access for required blood sampling
* Unable to attend all visits required by the protocol
* Female patients must be EXCLUDED if they are pregnant, breast feeding, planning to become pregnant during the study or using hormonal contraception as their only method of birth control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in Westhaven Scale | 4 weeks

SECONDARY OUTCOMES:
Efficacy: Change in Hepatic Encephalopathy Scoring Algorithm (HESA) | 4 weeks
Efficacy: Reduction of venous ammonia levels | 4 weeks
Efficacy: Serum bile acids and amino acid profile | 4 weeks
Efficacy: Reduction in itching (visual analog scale) | 4 weeks
Efficacy: Presence or absence of asterixis | 4 weeks
Safety: Clinical laboratory tests | 4 weeks
Safety: Physical examination, vital signs (blood pressure, heart rate, respiration rate, body temperature) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pockros, MD, Principal Investigator — Scripps Clinic
Locations (17):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - Scripps Clinic, San Diego, California
  - Veterans Medical Center San Diego, San Diego, California
  - Washington Hospital Center - MedStar Research Institute, Washington D.C., District of Columbia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Massachusetts Medical School, Worchester, Massachusetts
  - Weill Medical College of Cornell, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - Baylor University Medical Center, Houston, Texas
  - St. Luke's Advanced Liver Therapies / St. Luke's Texas Liver Coalition - Baylor College of Medicine, Houston, Texas
  - Metropolitan Research, Fairfax, Virginia
  - McGuire VA Medical Center, Richmond, Virginia